CLINICAL TRIAL: NCT01182259
Title: The Incidence and Risk Factors of Side Effects During the Initial Phase of Rifater Therapy - a Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: E-DA Hospital (Other)
Other Study IDs: JTWu002
Record Dates: First submitted 2010-08-13; First posted 2010-08-16 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Tuberculosis remains one of the largest health problems in the world today. Multidrug therapy is necessary to cure tuberculosis patients and to prevent the selection of drug-resistant mutants, however, which may increase the incidence of side effects during the course of treatment. These side effects may be mild as well as fatal. A severe side effect against one of the anti-TB drugs, which influences drug compliance, may lead to the discontinuation of that drug. At the same time, the risk of treatment failure and relapse are higher. Therefore monitoring the rate of anti-TB drugs induced adverse effects and the related risk factors is crucial. Awareness of the risk groups may decrease the incidence of serious drug-related side effects and medical cost.

The fixed-dose combinations (FDCs) of tablets against tuberculosis is now being recommended by WHO, which simplify the prescription of drugs and prevent the development of drug resistance. However, the FDC regimen is not consistent with the dosages that are usually given, the higher risk of drug toxicity and adverse reactions should be considered. To our knowledge, there was no report to assess the adverse effects of FDC anti-TB drugs in Taiwan. The aim of the present study is to investigate the current incidence of side effects and the risk factors related to FDC drugs for side effects during the initial phase of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed pulmonary TB and extrapulmonary TB patients
2. No previous anti-TB drugs treatment
3. Age more than 18years old

Exclusion Criteria:

1. Expected life < 6months
2. Baseline AST and ALT > 3 fold upper limit of normal (ULN) or total bilirubin>2mg/dl
3. Age less than 18years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed TB patient in E-DA hospital
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-10

CONTACTS AND LOCATIONS:
Locations (1):
- E-DA hospital, Kaohsiung City, Taiwan